CLINICAL TRIAL: NCT05478395
Title: Correlation of Mukbang Video Watching Behavior,Internet Addition and Mental Health Among Adolescent and Youth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Other Study IDs: L2022SYSU-HL-027
Record Dates: First submitted 2022-07-27; First posted 2022-07-28 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Mukbang
Keywords: Mukbang; Mental Health; Internet Addiction
MeSH Terms: conditions — Psychological Well-Being; Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed adolescents and young adults: 1. Internet users aged 14-35;
  2. Be able to read and communicate in Chinese.
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — Participants will be asked to respond to the demographic information，the Depression Anxiety Stress Scale（DASS-21）and the Internet Addiction Test（IAT）.

SUMMARY:
The mental health and Internet addiction problems of adolescents and youth can not be ignored and need to be solved urgently. The behavior of watching "Mukbang" videos may be in a mediating position between the two, and its specific effects and mechanisms are still unclear. Based on the theory of use and satisfaction, this study will further explore the interactive relationship between "Mukbang" and mental health and Internet addiction from the perspective of adolescents and young Internet users. Thereby enriching research paths in related fields and providing theoretical basis for clinical mental health guidance or intervention.

DETAILED DESCRIPTION:
Adolescence and Youth is a critical period for psychological quality training and personality shaping, and their mental health has always been the focus of health management for this population. With the rapid development of short videos and self-media, watching "Mukbang" is a behavioral way for these people to relieve anxiety, depression and other mental health problems. But watching "Mukbang" behaviors may have Internet addiction, and there is a high comorbidity rate between Internet addiction and mental health disorders. "Mukbang" is a newly developed online entertainment method. Its helpfulness in reducing psychological stress, relieving depression and other negative emotions, and the mechanism of action that aggravates the risk of Internet addiction is unknown. At present, the new crown epidemic is spreading all over the world, and the stress reactions such as fear, anxiety, sadness and anger brought to teenagers and young people will induce more psychological problems; and closed management has greatly increased the risk of such people. Internet addiction time, the detection rate of Internet addiction has also greatly increased, resulting in a serious vicious circle. Based on the theory of use and satisfaction, this research will adopt an exploratory time-series mixed design. First, qualitative research is used to explore the possible reasons and related experience of adolescents and young people watching "eating and broadcasting"; Potential related variables and quantitative indicators of watching "eating and broadcasting" behavior, further verify the correlation between "eating and broadcasting" behavior, Internet addiction and mental health; and explore the role of "eating and broadcasting" video watching behavior in mental health and Internet addiction. mediation between them. It provides a theoretical basis for promoting the healthy and psychological development of adolescents and young people, standardizing the management of "eating and broadcasting" videos, and correcting the correct guidance for preventing addiction to the Internet.

ELIGIBILITY:
Inclusion Criteria:

* Internet users aged 14-35；
* Be able to read and communicate in Chinese.

Exclusion Criteria:

* Those who cannot complete communication due to serious mental or physical diseases such as deafness, unclear consciousness caused by mental illness, etc.

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents and young adults
Sampling Method: Non-Probability Sample
Enrollment: 1035 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Features of Watching "Mukbang" Videos | Baseline
  The"Mukbang" watching features will be assessed by a questionnaire designed by the researcher and recorded by the subjects themselves, including watching time, watching rate, watching preferences and watching experience.
Mental Health | Baseline
  The mental health status will be assessed by the Depression Anxiety Stress Scale（DASS-21），4-point Likert rating scale, which contains 21 items to describe personal recent negative emotional experience. The full scale consists of three subscales of depression, anxiety and stress, each of which contains 7 items.
Internet Addiction | Baseline
  The Internet addiction risk will be assessed by the Chinese version of Young's self-rating Internet addiction scale，a total of 20 items. Each item used a 5-point Likert scale(1=rarely, 2=occasionally, 3=sometimes, 5=always), and the total score ranged from 20 to 100. The higher the score, the more serious the risk of Internet addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No